CLINICAL TRIAL: NCT03909568
Title: A Randomised Controlled Trial to Assess the Alveolar Bone Height Distal to Lower Second Molar Following Either Coronectomy or Extraction of the Adjacent Impacted Lower Third Molar
Brief Title: Bone Height and Extractions Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 249253
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-04

CONDITIONS: Alveolar Bone Loss; Periodontal Attachment Loss; Periodontal Pocket
MeSH Terms: conditions — Alveolar Bone Loss; Periodontal Attachment Loss; Periodontal Pocket

STUDY DESIGN:
Intervention Model Description: Split-mouth
Masking Description: Patients will be initially masked to which treatment is performed on each side, but will be notified at the follow-up appointment. In addition, the outcomes assessor carrying out the periodontal measurements (clinical attachment level and probing depths), will be unaware which treatment will be performed. The same surgical flap designs will be used for the treatment of both the right and left third molars, regardless of whether a coronectomy or extraction is carried out, and therefore the patient and clinician should be unable to differentiate between the procedures performed. Intervention will only be revealed to care provider once surgical flaps have been raised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Third molar surgery (Experimental): Split mouth comparison of effect of complete third molar removal vs coronectomy of contralateral third molar
  Interventions: Procedure: Third molar surgery

INTERVENTIONS:
Procedure: Third molar surgery — Comparing complete removal of third molar with removal of crown only on contralateral side

SUMMARY:
A coronectomy is often chosen over complete extraction of a lower third molar when the tooth appears to be in close proximity to the inferior dental (ID) canal, as assessed on a plain radiograph or a cone beam computer tomograph (CBCT). Following a coronectomy, the roots of the third molar may migrate in a coronal direction. This effect, along with the bone-preserving technique of a coronectomy over extraction, may provide increased bone height distal to the lower second molars, when compared to extraction. Partially erupted lower third molars, specifically those with mesio-angular impactions, are commonly associated with reduced bone height distal to lower second molars, and cause damage to the periodontal support of these neighboring teeth. It is assumed that maintenance of the impacted third molars or extraction of these teeth may compromise the periodontal status of the lower second molars. This study will investigate if coronectomy improves the bone levels, and therefore the periodontal status, of lower second molars, and may propose an indication for a coronectomy regardless of the proximity of the tooth to the ID canal.

Coronectomies were first proposed as a treatment option just over thirty years ago, but there are very few long-term studies on the procedure reported in the literature. To the best of the investigator's knowledge, this will be the first randomised controlled trial comparing the bone height distal to the lower second molar following a coronectomy or extraction of the lower third molar.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring extraction of both lower third molars
* Both lower third molars to have mesio-angular impa
* ctions, as assessed by location of the contact point between the crown of the third molar and the cemento-enamel junction (CEJ) of the second molar and the angulation of the third molar
* Both lower third molars must lie above or clear of the ID canal as assessed on a plain radiograph or CBCT
* Presence of lower second molars
* Patients must be ≥18yrs old
* Patients willing to attend follow up appointments

Exclusion Criteria:

* Lower third molars with caries, periapical pathology or associated lesions such as cysts
* Patients who are immunocompromised, have a history of or due to have head and neck radiotherapy, chemotherapy, have previously been given or due to start intravenous bisphosphonates
* Smokers (>5 cigarettes/day)
* Patients involved in current research or have recently been involved with research prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Linear bone height distal to lower second molar tooth | Six months surgical intervention
  Assessed by comparison of periapical radiographs pre- and post-intervention

IPD SHARING:
Plan to Share IPD: No